CLINICAL TRIAL: NCT02424773
Title: Oxygen Therapy During Acute Respiratory Failure in Immuno-compromised Patients
Acronym: RESPIR-OH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K101201
Record Dates: First submitted 2015-04-20; First posted 2015-04-23 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2015-04

CONDITIONS: Acute Respiratory Failure; Immunocompromised Host; High Flow Oxygen Cannula
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Venturi group (Active Comparator): Venturi group : Oxygen is delivered using oxygen Venturi mask FiO2 is started at 60% (15l/min) and modified to maintain SpO2 over 94%.
  Interventions: Device: Venturi mask; Drug: Oxygen
- HFNC group (Experimental): HFNC group : Oxygen is delivered using HFNC. HFNC is started with FIO2 =1 and modified to maintain SpO2 over 94%, flow is settled at 40-50l/min.
  Interventions: Device: High Flow Nasal Canula (HFNC); Drug: Oxygen

INTERVENTIONS:
Device: High Flow Nasal Canula (HFNC)
  Arms: HFNC group
Device: Venturi mask
  Arms: Venturi group
Drug: Oxygen

SUMMARY:
In immunocompromised patients, Acute Respiratory Failure (ARF) is associated with a high case-fatality, particularly when invasive Mechanical Ventilation (MV) is required. In the most hypoxemic patients, oxygen administration through High Flow Nasal Cannula (HFNC) has been reported as an alternative to the venturi mask. The aim of this study is to compare HFNC and venturi mask on early respiratory deterioration and patient's comfort in that setting. The investigators planned a prospective randomized study in 4 Intensive Care Units (ICUs). As respiratory deterioration occurs early after ICU admission, patients are randomized to receive two hours of oxygen therapy either through HFNC or venturi mask. The primary endpoint is defined as the need for invasive or noninvasive MV in the 2-hour period. Secondary endpoints include comfort, dyspnea and thirst.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years.
* Admission to ICU for ARF. ARF was defined with the need of oxygen over 6l/min to maintain SpO2 over 95% or symptom of respiratory distress (intercostal recession or tachypnea >30/min or dyspnea at rest).
* Immunosuppression. Immunosuppressed conditions were solid tumor, hematological malignancy, steroid treatment or other immunosuppressive treatment, or HIV infection.

Exclusion Criteria:

* Hypercapnia (above 47 mmHg)
* Chronic respiratory failure
* Previous mechanical ventilation in the days before admission
* Need of immediate NIV or intubation
* Refusal
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-11; Primary Completion 2014-11 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Oxygenation failure | 2 hours
  Oxygenation failure is defined with the need of invasive Mechanical Ventilation or Non invasive ventilation during the two hours study period

SECONDARY OUTCOMES:
comfort (0-10 Visual analog Scale) | 1 hour
  0-10 Visual analog Scale
comfort (0-10 Visual analog Scale) | 2 hours
  0-10 Visual analog Scale
dyspnea (0-10 Visual analog Scale) | 1 hour
  0-10 Visual analog Scale
dyspnea (0-10 Visual analog Scale) | 2 hour
  0-10 Visual analog Scale
thirst (0-10 Visual analog Scale) | 1 hour
  0-10 Visual analog Scale
thirst (0-10 Visual analog Scale) | 2 hour
  0-10 Visual analog Scale

CONTACTS AND LOCATIONS:
Overall Officials: Sophie COURTIAL DESTEMBERT, Study Director — DRCD APHP Paris

REFERENCES:
- [Result] Lemiale V, Mokart D, Mayaux J, Lambert J, Rabbat A, Demoule A, Azoulay E. The effects of a 2-h trial of high-flow oxygen by nasal cannula versus Venturi mask in immunocompromised patients with hypoxemic acute respiratory failure: a multicenter randomized trial. Crit Care. 2015 Nov 2;19:380. doi: 10.1186/s13054-015-1097-0. PMID 26521922